CLINICAL TRIAL: NCT02029300
Title: A Randomized Comparison of Nasal Versus Oral Fiberoptic Intubation in Children Less Than Two Years of Age
Brief Title: A Comparison of Nasal Versus Oral Fiberoptic Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Pediatric Anesthesiologist, Associate Professor of Anesthesiology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-15520
Record Dates: First submitted 2013-11-07; First posted 2014-01-07 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Tracheal Intubation
Keywords: pediatrics; fiberoptic intubation; oral intubation; nasal intubation; children under the age of 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Route (Other): The nasal route will be when the airway is acquired and secured with a fiberoptic bronchoscope through one of the nares.
  Interventions: Other: Fiberoptic Intubation through the nasal route
- Oral Route (Other): The oral route will be when the airway is acquired and secured with a fiberoptic bronchoscope through the patient's mouth.
  Interventions: Other: Fiberoptic intubation through the oral route

INTERVENTIONS:
Other: Fiberoptic Intubation through the nasal route
  Arms: Nasal Route
Other: Fiberoptic intubation through the oral route
  Arms: Oral Route

SUMMARY:
There are two routes in which a fiberoptic intubation can be performed - oral and nasal. In general, nasal intubation by any conventional method may be the preferred choice for certain procedures such as intra-oral surgeries, or for anatomical reasons such as limited mouth opening. If nasal intubation is not indicated or preferred, then oral intubation is usually performed.

This study is looking to explore whether or not the nasal route significantly improves the ease and time for successful fiberoptic intubation compared to the oral route in children less than or equal to 2 years of age. This study will also examine if operator experience influence time to tracheal intubation with either route?

The investigators hypothesize that the nasal route of fiberoptic intubation will be faster than the oral route, for both the trainee and the expert, and that there will be minimal differences between experts and trainees with nasal fiberoptic intubation.

DETAILED DESCRIPTION:
The goal of this prospective randomized study is to compare the effect of nasal fiberoptic intubation versus oral fiberoptic intubation in children less than 2 years of age. Other factors that will be assesed include operator experience, the ease and time for fiberoptic grade of laryngeal view, time for fiberoptic tracheal intubation, and complications.

This study is looking to explore whether or not the nasal route significantly improves the ease and time for successful fiberoptic intubation compared to the oral route in children less than or equal to 2 years of age. While also asking, will operator experience influence time to tracheal intubation with either route?

The investigators hypothesize that the nasal route fiberoptic intubation will be faster than the oral route, for both the trainee and the expert, and that there will be minimal differences between experts and trainees with nasal fiberoptic intubation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children ASA I to III
* Patients less than or equal to 2 years of age
* Patients with scheduled surgeries in which endotracheal intubation is part of their general anesthetic plan

Exclusion Criteria:

* Children with ASA IV or V
* Children with active respiratory infection, pulmonary disease, a known history of difficult mask ventilation, high suspicion of difficult airway (secondary to congenital syndromes for example), and significant airway abnormalities

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time to fiberoptic intubation | From disconnection of oxygen to reconnection of oxygen during tracheal intubation

OTHER OUTCOMES:
Time to first glottic view | during tracheal intubation
  This will be measuring the time it takes the anesthesiologist to have the first glottic view.
Time to carinal view | during tracheal intubation
  This is the time it will take the anesthesiologist to the first carinal view.
Time to successful intubation | during tracheal intubation
  This will measure the entire time period it takes for the ansthesiologist to intubate the patient.
Complications | From the beginning to the end of intubation, and after the surgery up to 24 hours post-op
  Complications will be recorded and defined as follows:
  * laryngospasm: clinical evidence of inability to ventilate
  * bronchospasm: bilaterally inspiratory and expiratory wheezing along with potential desaturations and changes in capnogram morphology
  * desaturation: SpO2 (blood oxygen saturation) below 90% at any time during the case

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Lurie Childrens Hospital
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Wheeler M, Roth AG, Dsida RM, Rae B, Seshadri R, Sullivan CL, Heffner CL, Cote CJ. Teaching residents pediatric fiberoptic intubation of the trachea: traditional fiberscope with an eyepiece versus a video-assisted technique using a fiberscope with an integrated camera. Anesthesiology. 2004 Oct;101(4):842-6. doi: 10.1097/00000542-200410000-00007. PMID 15448515
- [Derived] Jagannathan N, Sequera-Ramos L, Sohn L, Huang A, Sawardekar A, Wasson N, Miriyala A, De Oliveira GS. Randomized comparison of experts and trainees with nasal and oral fibreoptic intubation in children less than 2 yr of age. Br J Anaesth. 2015 Feb;114(2):290-6. doi: 10.1093/bja/aeu370. Epub 2014 Nov 5. PMID 25377166